CLINICAL TRIAL: NCT00372788
Title: A Phase II, Open, Randomised Study to Assess the Efficacy and Safety of AZD6244 Versus Pemetrexed (Alimta®) in Patients With Non-small Cell Lung Cancer, Who Have Failed One or Two Prior Chemotherapy Regimen
Brief Title: AZD6244 Versus Pemetrexed (Alimta®) in Patients With Non-small Cell Lung Cancer, Who Have Failed One or Two Prior Chemotherapy Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00012
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Advanced Non-Small Cell Lung Cancer; AZD6244
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — AZD 6244; Pemetrexed

ARMS (2):
- 1 (Active Comparator): Pemetrexed
  Interventions: Drug: Pemetrexed
- 2 (Experimental): AZD6244
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — oral vial
  Other Names: ARRY-142886
  Arms: 2
Drug: Pemetrexed — oral
  Other Names: Alimta®
  Arms: 1

SUMMARY:
The purpose of this study is to assess the effect and safety of AZD6244(ARRY-142886)versus pemetrexed in the second or third line treatment of advanced Non-Small Cell Lung Cancer. Following baseline assessments, a minimum of 64 patients in approximately 5-6 centers from the US will be treated with either AZD6244 or pemetrexed. Treatment will be continued for as long as patients receive clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-small cell lung cancer
* Previously received one or two chemotherapeutic treatments

Exclusion Criteria:

* Previous therapy with MEK inhibitor or pemetrexed
* Any recent surgery, unhealed surgical incision or severe condition such as uncontrolled cardiac disease or chronic gastrointestinal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assess tumor growth | assessed every 12 weeks

SECONDARY OUTCOMES:
Assess safety and tolerability of AZD6244 | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Emerging Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (8):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, Ann Arbor, Michigan
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Research Site, Cluj-Napoca, Romania

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1173&filename=CSR-D1532C00012.pdf
- See also: CSR-D1532C00012.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1173&filename=CSR-D1532C00012.pdf